CLINICAL TRIAL: NCT06917313
Title: A Randomized Phase II Study to Evaluate the Efficacy of Fezolinetant in Reducing Vasomotor Symptoms in Women With Breast Cancer on Endocrine Therapy
Brief Title: FLASH-Breast: Evaluating the Efficacy of Fezolinetant in Reducing Vasomotor Symptoms in Women With Breast Cancer on Endocrine Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Maryam Lustberg, Professor of Internal Medicine, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000037181
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: adjuvant endocrine therapy; vasomotor symptoms; tamoxifen; aromatase
MeSH Terms: interventions — fezolinetant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fezolinetant (Active Comparator): Fezolinetant is an oral medication, and the first neurokinin 3 (NK3) receptor antagonist approved by the FDA in May 2023 for treatment of moderate to severe hot flashes due to menopause. It blocks the activities of the NK3 receptor which is involved in the brain's regulation of body temperature.
  Interventions: Drug: Fezolinetant
- Placebo (Placebo Comparator): Patients will be given placebo tablets to compare to active comparator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fezolinetant — 45 mg tablets, administered orally once daily with or without food, to be taken throughout the entire study phase, i.e. 12 weeks
  Arms: Fezolinetant
Drug: Placebo — 45 mg tablets, administered orally once daily with or without food, to be taken throughout the entire study phase, i.e. 12 weeks
  Arms: Placebo

SUMMARY:
This is a phase II, randomized, double-blinded, placebo-controlled trial designed to evaluate the efficacy of fezolinetant (45 mg a day) vs. placebo in reducing moderate to severe vasomotor symptoms (VMS) in breast cancer survivors on endocrine therapy (tamoxifen, aromatase inhibitors). The trial will proceed in a single stage, and the total of 92 participants will be randomized in 1:1 fashion to fezolinetant or placebo arm respectively.

DETAILED DESCRIPTION:
This is a phase II, randomized, double-blinded, placebo-controlled trial designed to evaluate the efficacy of fezolinetant (45 mg a day) vs. placebo in reducing moderate to severe vasomotor symptoms (VMS) in breast cancer survivors on endocrine therapy (tamoxifen, aromatase inhibitors). The trial will proceed in a single stage, and the total of 92 participants will be randomized in 1:1 fashion to fezolinetant or placebo arm respectively. After the 7-14-day screening period when all the baseline, pre-treatment measures will be collected, we will record daily data on frequency and severity of VMS and calculate weekly averages of both metrics. After the 12 weeks treatment period, formal efficacy analysis will be conducted and the treatment with fezolinetant will be deemed efficacious if the final weekly average of daily frequency of VMS will be significantly reduced compared to the 'week12 - baseline' difference of the placebo arm. Upon conclusion of the formal 12-week treatment assignment, once VMS final assessment has been recorded, we will unblind the study participants to their treatment assignment. Participants will be then allowed to cross over shall they choose to do so. Due to the vast availability of safety and efficacy data in general population, we did not include interim efficacy/futility or safety analysis.

Our hypothesis is that neurokinin blockade by fezolinetant will significantly reduce vasomotor symptoms in breast cancer survivors on endocrine therapy (tamoxifen or aromatase-inhibitor) measured by mean change in frequency of moderate to severe VMS based on patient-reported data from baseline to 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

Women with diagnosed, histologically confirmed, clinical stage I-III, HR+ invasive breast cancer as defined by ASCO CAP guidelines for whom adjuvant endocrine therapy would be indicated.

BMI of 18-40 kg/m2

Age 40-65

Currently on endocrine therapy (tamoxifen or aromatase inhibitors)

Willing and able to provide written informed consent/assent for the trial.

Postmenopausal as defined by spontaneous amenorrhea for at least 12 consecutive months, spontaneous amenorrhea for at least 6 months with biochemical criteria or menopause (FSH > 40 IU/L), or bilateral oophorectomy for at least 6 weeks before the screening visit, or if premenopausal chemically suppressed by GnRH agonist therapy with ultrasensitive estradiol level <10.

On endocrine therapy for a minimum of 3 months and has planned duration of 12 weeks left in the treatment regimen.

Experiencing an average of seven or more moderate to severe hot flashes per day over a 7-day period as documented by Symptom Diary during the Screening Period and seeking treatment or relief for VMS.

Able to swallow oral formulation of the study agent.

Exclusion Criteria:

Participants who have a diagnosis of stage IV metastatic disease

Receiving any other cancer treatment other than endocrine therapy. This includes chemotherapy, targeted therapies, and immunotherapy.

Receiving cytochrome CYP1A2 inhibitors

Participants who have received any treatment for vasomotor symptoms (prescription, over the counter, or herbal) for the last 28 days.

Pregnant or lactating patients

Active liver disease, jaundice, or elevated liver aminotransferases (ALT or AST) >2x ULN, or elevated total bilirubin, OR elevated direct bilirubin, or elevated INR, or elevated alkaline phosphatase >2x ULN

Creatinine > 1.5 times upper limit of normal; or estimated GFR ≤ 30 mL/min per 1.73 m2 at screening.

Judgement by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Frequency of moderate/severe VMS at 12 weeks of treatment with fezolinetant vs. placebo | Baseline to 12 weeks
  To evaluate the mean change reduction in frequency of moderate/severe VMS at 12 weeks of treatment with fezolinetant vs. placebo in breast cancer survivors on endocrine therapy (tamoxifen or aromatase inhibitors).

SECONDARY OUTCOMES:
Efficacy of fezolinetant vs. placebo in reducing the mean daily frequency of moderate/severe VMS | At week 4, after treatment initiation
  To evaluate the efficacy of fezolinetant vs. placebo in reducing the mean daily frequency of moderate/severe VMS
Regression of mean daily frequency of moderate/severe VMS average | Study duration: weeks 0-12
  To evaluate treatment activity among breast cancer survivors treated with fezolinetant vs placebo over the entire course of the study duration - measure by regression of mean daily frequency of moderate/severe VMS average every week of treatment (weeks 0-12)
Change in global quality of life using Functional Assessment of Cancer Therapy - Breast, Endocrine Therapy Symptoms (FACT-B ES) | Baseline to week 12
  To evaluate the difference in global quality of life in breast cancer survivors treated with fezolinetant vs placebo using FACT-B ES. The total score range is 0 to 164, with higher scores indicating better quality of life
Differences in sleep quality using PROMIS Sleep Disturbance-Short Form 8b (PROMIS SD SF 8b) | Baseline, week 4 and week 12
  To evaluate the differences in sleep quality in breast cancer survivors' treatment with fezolinetant vs placebo using patient-reported outcomes measurement information System Sleep Disturbance - Short Form 8b (PROMIS SD SF 8b. Total score is calculated by summing the items (range: 8-40), with a higher score meaning more disturbed sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Lustberg, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No